CLINICAL TRIAL: NCT05274984
Title: Lidocaine Continuous Infusion for ERCP Procedures: a Prospective, Randomized, Double-blinded, Controlled Trial
Brief Title: Lidocaine Infusion for Propofol Dose Reduction in ERCP Procedure
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Breazu Caius Mihai, Assistant Professor MD PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIP
Record Dates: First submitted 2022-02-17; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Sedation
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to controll group or lidocaine group. Participants of control group are given placebo while participants of lidocaine group are given lidocaine.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, endoscopist, anesthetist, and data collection observers were all blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Placebo (Placebo Comparator): the control group will be given the same volume of saline as the experimental group
  Interventions: Drug: Placebo
- Group Lidocaine (Active Comparator): the experimental group will be given l-1.5mg lidocaine and then 2mg/kg/h
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Placebo — the control group will be given the same volume of saline.
  Arms: Group Placebo
Drug: Lidocaine — the experimental group will be given 1.5mg/kg lidocaine and then 2mg/kg/h
  Arms: Group Lidocaine

SUMMARY:
This study aims to investigate the dose reduction of propofol if associated with continuous infusion of lidocaine during ERCP procedures in patients over 65 years old.

DETAILED DESCRIPTION:
The primary aim of this study was to evaluate the effect of continuous infusion of lidocaine on propofol consumption in older patients having ERCP sedation. Secondary outcomes were to evaluate patient adverse events, sedation quality and satisfaction of the patient and the endoscopist, postprocedural pain, and sedation-related time.For this the investigators randomised patients into 2 groups: Group Lidocaine received 1,5 mg/kg lidocaine 1% 10 min before procedure and then 2 mg/kg/h continuous infusion of lidocaine 1%, whereas the Group Control received an equal volume of saline solution, which could not be visually identified from lidocaine by the blinded anaesthesiologist. All patients received propofol bolus dose of 1mg/kg than 10-20 mg iv boluses during the procedure guided by capnograph monitoring and the patient's grimace, mobility, hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

* 65-85 years old
* physical status ASA I, II, III,
* ERCP scheduled

Exclusion Criteria:

* ASA IV or higher
* severe renal, cardiac or liver failure,
* allergy to lidocaine,
* patients weighing less than 40 kg,
* inability to give informed consent

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-03-03 (Estimated); Study Completion 2022-04-03 (Estimated)

PRIMARY OUTCOMES:
Propofol consumption between the 2 groups | During ERCP procedure
  To evaluate propofol consumption by recording total dose of propofol(mg) during ERCP procedure between the 2 groups.

SECONDARY OUTCOMES:
Safety assessed by the rate of hypoxia during the procedure | During ERCP procedure
  Recording the number of hypoxia episodes, defined as peripheral oxygen saturation <94% for >30 seconds during ERCP procedure between the 2 groups.
Safety assessed by the rate of involuntary movement during the procedure | During ERCP procedure
  Number of involuntary movements, defined as unconscious movements requiring restraint of patients during ERCP procedure between the 2 groups
Lidocaine | During ERCP procedure
  Asses the total dose of lidocaine (mg) used in GROUP Lidocaine during ERCP procedure
Endoscopist satisfaction between 2 groups | After ERCP procedure
  The endoscopists satisfaction score to be assessed on a 1-4 VAS after the procedure ( 1-poor, 2-moderate, 3-good, 4-excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ionescu, MD PhD, Study Chair — UMF Iuliu Hatieganu Cluj-Napoca
Locations (1):
- Regional Institute of Gastroenterology and Hepatology "Prof.dr.Octavian Fodor", Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No